CLINICAL TRIAL: NCT05181592
Title: A Phase IIIb, Open-label, Single Arm Study to Evaluate the Efficacy and Safety of Luspatercept in Patients With Lower-risk MDS and Ring-sideroblastic Phenotype (MDS-RS)
Brief Title: Assessment of Effectiveness and Safety of Luspatercept in Patients Suffering From Lower-risk Myelodysplastic Syndrome.
Acronym: LUSPLUS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GWT-TUD GmbH (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUSPLUS
Record Dates: First submitted 2021-12-02; First posted 2022-01-06 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS; Luspatercept; myelodysplastic syndrome; ring-sideroblastic phenotype; MDS-RS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — luspatercept

STUDY DESIGN:
Intervention Model Description: International, multicenter, non-comparative, open-label, single arm study
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Luspatercept (single arm) (Experimental): open-label, single-arm
  Interventions: Drug: Luspatercept

INTERVENTIONS:
Drug: Luspatercept — Once 1.75 mg/kg on Day 1 of each 21-day cycle for 24 weeks (9 cycles)
  Other Names: Reblozyl

SUMMARY:
A phase IIIb, open-label, single arm study to evaluate the efficacy and safety of luspatercept in patients with lower-risk MDS and ring-sideroblastic phenotype (MDS-RS)

DETAILED DESCRIPTION:
This is a phase IIIb, single arm, multicenter study to further explore the efficacy and safety of luspatercept in subjects with anemia due to IPSS-R very low-, low-, or intermediate-risk MDS with RS who require RBC transfusions. The study will consist of a screening period, a treatment period (primary phase and extension phase), and a posttreatment follow-up period.

The study will involve study sites in Germany, France, Austria and Switzerland. It is planned to include 70 patients to receive treatment with luspatercept to end up with 64 evaluable subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years of age or older at the time of signing the informed consent form (ICF)
2. Subject is able to understand and voluntarily sign the ICF prior to any study-related assessments/procedures being conducted
3. Subject has documented diagnosis of MDS according to WHO classification that meets IPSS-R classification[3] of very low-, low-, or intermediate-risk disease, and the following:

   * Ring sideroblasts (RS) ≥ 15% of erythroid precursors in bone marrow or ≥ 5% if SF3B1 mutation is present
   * Less than 5% blasts in bone marrow
   * Peripheral blood white blood cell (WBC) count < 13,000/μL
4. Subject must be one of the following:

   * Refractory to prior ESA treatment: Documentation of non-response or response that was no longer maintained to prior ESA-containing regimen, either as a single agent or in combination (e.g. with granulocyte colony-stimulating factor [G-CSF]). The ESA regimen must be either:

     * Recombinant human erythropoietin ≥ 40,000 IU/week for at least 8 weeks (=doses) or equivalent; or
     * Darbepoetin-α ≥ 500 μg q3w for at least 4 doses or equivalent
   * Intolerant to prior ESA treatment: Documentation of discontinuation of prior ESA containing regimen, either as a single agent or in combination (e.g. with G-CSF), at any time after introduction due to intolerance or an adverse event (AE)
   * ESA ineligible: Low chance of response to ESA based on endogenous serum erythropoietin (EPO) level > 200 U/L for subjects not previously treated with ESAs
   * Refractory to- /relapsed after prior HMA treatment1: Treatment failure/relapse after at least six (azacitidine) or four (decitabine) 4-week treatment cycles except for del(5q) MDS
   * Refractory to- /relapsed after prior lenalidomide treatment1 except for del(5q) MDS
5. If previously treated with ESAs or G-CSF/granulocyte-macrophage colony-stimulating factor (GM-CSF), both agents must be discontinued ≥ 4 weeks prior to the date of starting treatment with the Investigational medicinal Product (IMP) in this study
6. Required RBC transfusions, as documented by the following criteria:

   * Average transfusion requirement of ≥ 2 units/8 weeks of packed RBCs confirmed for a minimum period of 16 weeks immediately preceding start of treatment with IMP
   * Hemoglobin (Hb) levels at the time of or within 7 days prior to administration of an RBC transfusion must be ≤ 10.0 g/dL in order for the transfusion to be counted towards meeting eligibility criteria. RBC transfusions administered when Hb levels are > 10 g/dL and/or RBC transfusions administered for elective surgery do not qualify as a required transfusion for the purpose of meeting eligibility criteria
   * No consecutive 56-day period that is RBC transfusion-free during the 16 weeks immediately prior to starting treatment with IMP
7. Eastern Cooperative Oncology Group (ECOG) score of 0, 1, or 2
8. A female of childbearing potential (FCBP) for this study is defined as a sexually mature woman who: (1) has not undergone a hysterectomy or bilateral oophorectomy; or (2) is not naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e. had menses at any time in the preceding 24 consecutive months). An FCBP participating in the study must:

   * Have 2 negative pregnancy tests as verified by the investigator prior to starting IMP (unless the screening pregnancy test is done within 72 hours of Cycle 1 Day 1). She must agree to ongoing pregnancy testing during the course of the study and after end of treatment (EOT).
   * If sexually active, agree to use, and be able to comply with, highly effective contraception** without interruption, 5 weeks prior to starting IMP, during treatment with IMP (including dose interruptions), and for 12 weeks after discontinuation of IMP. ** Highly effective contraception is defined in this protocol as the following (information also appears in the ICF): Hormonal contraception (e.g. birth control pills, injection, implant, transdermal patch, vaginal ring), intrauterine device, tubal ligation, or a partner with a vasectomy
9. Male subjects must agree to use a condom, defined as a male latex condom or nonlatex condom NOT made out of natural (animal) membrane (e.g. polyurethane), during sexual contact with a pregnant female or an FCBP while participating in the study, during dose interruptions, and for at least 12 weeks following IMP discontinuation, even if he has undergone a successful vasectomy
10. Subject is willing and able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

1. Prior therapy with disease modifying agents other than HMA or LEN for underlying MDS disease
2. Previously treated with either luspatercept or sotatercept
3. Secondary MDS, i.e. MDS that is known to have arisen as the result of chemical injury or treatment with chemotherapy and/or radiation for other diseases
4. Known clinically significant anemia due to iron, vitamin B12, or folate deficiencies, or autoimmune or hereditary hemolytic anemia, or gastrointestinal bleeding

   • Iron deficiency to be determined by local laboratory via serum ferritin ≤ 15 μg/L and additional testing if clinically indicated (e.g. calculated transferrin saturation [iron/total iron binding capacity ≤ 20%] or bone marrow aspirate stain for iron)
5. Prior allogeneic or autologous stem cell transplant
6. Known history of diagnosis of acute myeloid leukemia (AML)
7. Use of any of the following within 5 weeks prior to the first dose of the IMP in this study:

   * Anticancer cytotoxic chemotherapeutic agent or treatment
   * Corticosteroid, except for subjects on a stable or decreasing dose for ≥ 1 week prior to the first dose of IMP for medical conditions other than MDS ICT, except for subjects on a stable or decreasing dose for at least 8 weeks prior to the first dose of IMP
   * Other RBC hematopoietic growth factors (e.g. interleukin [IL]-3)
   * Investigational drug or device, or approved therapy for investigational use. If the half-life of the previous study drug is known, the use of it within 5 times the half-life prior to the first dose of IMP or within 5 weeks, whichever is longer, is excluded
8. Uncontrolled hypertension, defined as repeated elevations of diastolic blood pressure (DBP) ≥ 100 mmHg despite adequate treatment
9. Platelet count < 30,000/μL (30 × 109/L)
10. Estimated glomerular filtration rate or creatinine clearance < 40 mL/min
11. Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) or alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) ≥ 3.0 × upper limit of normal (ULN)
12. Total bilirubin ≥ 2.0 × ULN

    * Higher levels are acceptable if these can be attributed to active RBC precursor destruction within the bone marrow (i.e. ineffective erythropoiesis) or in the presence of known history of Gilbert Syndrome
    * Subjects are excluded if there is evidence of autoimmune hemolytic anemia manifested as a corrected reticulocyte count of > 2% with either a positive Coombs test or over 50% indirect bilirubin
13. Prior history of malignancies, other than MDS, unless the subject is free of the disease (including completion of any active or adjuvant treatment for prior malignancy) for ≥ 5 years. However, subjects with the following history/concurrent conditions are allowed:

    * Basal or squamous cell carcinoma of the skin
    * Carcinoma in situ of the cervix
    * Carcinoma in situ of the breast
    * Incidental histologic finding of prostate cancer (T1a or T1b using the tumor, nodes, metastasis clinical staging system)
14. Major surgery within 8 weeks prior to the first dose of IMP. Subjects must be completely recovered from any previous surgery prior to the first dose of IMP
15. History of stroke, deep venous thrombosis, pulmonary or arterial embolism within 6 months prior to the first dose of IMP
16. Pregnant or breast-feeding females
17. Myocardial infarction, uncontrolled angina, uncontrolled heart failure, or uncontrolled cardiac arrhythmia as determined by the investigator within 6 months prior to the first dose of IMP. Subjects with a known ejection fraction of ˂ 35%, confirmed by a local echocardiography or multigated acquisition scan (MUGA) performed within 6 months prior to the first dose of IMP, are excluded
18. Uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment), known human immunodeficiency virus (HIV), known evidence of active infectious hepatitis B, and/or known evidence of active hepatitis C
19. History of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the IMP
20. Subject is in custody by order of an authority or a court of law
21. Participation in another interventional clinical study within the last 3 months prior to signing the ICF or simultaneous participation in other clinical studies
22. Close affiliation with the investigator (e.g. a close relative) or persons working at the study site
23. Subject is an employee of the sponsor or involved Contract research Organization (CRO)
24. Criteria which in the opinion of the investigator preclude participation for scientific reasons, for reasons of compliance, or for reasons of the subject's safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
RBC-TI rate according to IWG 2018 modified criteria | from Week 1 through Week 24
  Evaluation of RBC-TI rate of luspatercept for the treatment of anemia due to IPSS-R very low-, low-, or intermediate-risk MDS in subjects with ring sideroblasts (RS) who require RBC transfusions (according to IWG 2018 criteria).

SECONDARY OUTCOMES:
RBC-TI rate according to IWG 2006 criteria | from Week 1 through Week 24 and through Week 52
  RBC-TI rates according to IWG 2006 criteria (Weeks 1-24 and Weeks 1-52) will be estimated and 97.5% lower confidence limit will be calculated analogously to the primary endpoint.
Median time to RBC-TI | Week 1 through Week 24 and through Week 52
  Time to RBC-TI will be summarized only for subjects who achieve RBC TI ≥ 8 weeks on treatment. It is defined as the time between start of IMP and the date onset of TI is first observed (i.e, Day 1 of 56 days without any RBC transfusions).
Median Duration of RBC-TI | Week 1 through Week 24 and through Week 52
  Duration of RBC-TI will be determined only for subjects who achieve RBC TI ≥ 8 weeks on treatment. Duration of RBC-TI is defined as the longest RBC-TI period during the treatment period. Duration of response starts at the date onset of TI is first observed (i.e, Day 1 of 56 days without any RBC transfusions). Transfusion response ends on the day of the first transfusion given after response is documented. Subjects who maintain RBC-TI through EOT will be censored at the date of treatment discontinuation or death, whichever occurs first.
Change in RBC units transfused | Week 9 through Week 24 and Week 37 through Week 52
  Total number of RBC units transfused over a fixed 16-weeks period (weeks 9-24; weeks 37-52) will be compared to the total number of RBC units transfused in the 16 weeks immediately prior to first IMP.
Proportion of subjects achieving mean Hb increase ≥ 1.0 g/dL | Week 1 through Week 24 and through Week 52
  Hemoglobin (Hb) increase ≥ 1.0 g/dL is defined as proportion of subjects with ≥ 1.0 g/dL Hb increase compared to baseline that is sustained over any consecutive 56-day period within a specified timeframe in the absence of RBC transfusions.
Proportion of subjects achieving modified hematologic improvement - erythroids (mHI-E) per IWG 2006 criteria | Week 1 through Week 24 and through Week 52
Proportion of subjects achieving hematologic improvement - neutrophils (HI-N) per IWG 2006 criteria | Week 1 through Week 24 and through Week 52
Proportion of subjects achieving hematologic improvement - platelets (HI-P) per IWG 2006 criteria | Week 1 through Week 24 and through Week 52
Mean change in serum ferritin | Week 9 through Week 24 and Week 37 through Week 52
  Mean change in serum ferritin (Week 9-24; Weeks 37-52) is calculated as the difference of post-baseline mean serum ferritin and baseline mean serum ferritin.
Mean Change in Mean Daily Dose of Iron Chelation Therapy (ICT) | Week 9 through Week 24 and Week 37 through Week 52
  The change in daily dose for each subject is calculated as the difference of post-baseline mean daily dose and baseline mean daily dose.
Proportion of subjects with progression to AML (acute myeloid leukemia) | Week 1 to Week 52
  Time to progression to AML is defined as the time between baseline (day1 of IMP administration) and first diagnosis of AML as per WHO classification of ≥ 20% blasts in peripheral blood or bone marrow.
Overall survival | Week 1 to Week 52
  Overall survival (OS) is defined as the time between start of IMP and death.
Change in PRO | Week 1 to Week 52 and to EOT
  In order to evaluate the Change in PRO questionnaires (from Week 1 to Week 52 and to EOT) utilizing EORTC QLQ-C30, changes from baseline in overall score and sub-scores will be calculated.
Change in PerfO | Week 1 to Week 52 and to EOT
  In order to evaluate the Change in PerfO questionnaires (from Week 1 to Week 52 and to EOT) utilizing "Timed Up and Gotest" (TUG), changes from baseline in overall score and sub-scores will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Götze, Prof., Principal Investigator — Klinikum rechts der Isar der Technischen Universität München
Locations (13):
- Austria (2):
  - Medizinische Universität Innsbruck, Innsbruck
  - Medizinische Universität Wien, Vienna
- Germany (2):
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum rechts der Isar, München
- Spain (6):
  - Institut Català d' Oncologia de Badalona, Badalona
  - Hospital Vall d´Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - University Hospital of Salamanca, Salamanca
  - Hospital Universitario y Politecnico La Fe de Valencia, Valencia
- Switzerland (3):
  - Universitätsspital Basel, Basel
  - Clinica di Ematologia Istituto oncologico della Svizzera Italiana, Bellinzona
  - Universitätsklinik für Hämatologie und Hämatologisches Zentrallabor, Bern

IPD SHARING:
Plan to Share IPD: No